CLINICAL TRIAL: NCT00161746
Title: Multicentre Randomized Double-Blind Phase II/III Study on the Safety and Immunogenicity of Three Vaccinations With TICOVAC in Two Dosages in Healthy Children Aged Between Six Months and Three Years
Brief Title: Safety and Immunogenicity Study of 3 Vaccinations With TICOVAC in 2 Dosages in Healthy Children Aged Between 6 Months and 3 Years
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 146A
Record Dates: First submitted 2005-09-08; First posted 2005-09-13 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Encephalitis, Tick-borne
Keywords: Tick-Borne Encephalitis
MeSH Terms: conditions — Encephalitis, Tick-Borne | interventions — Vaccines

INTERVENTIONS:
Biological: Tick-Borne Encephalitis (TBE) Vaccine (Inactivated)

SUMMARY:
The purpose of this study is to evaluate a) whether the seroconversion rates in children are equivalent after two and/or three partial vaccinations with TICOVAC 0.25 mL and TICOVAC 0.5 mL, and b) whether there is a difference in terms of safety between the two products.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children aged between 6 and 47 months
* No history of any previous TBE vaccination
* Clinically healthy
* Informed consent provided by the parents

Exclusion Criteria:

* History of allergic reactions, in particular allergic reactions to one of the components of the vaccine
* Suffering from a disease that cannot be effectively treated or stabilised
* Suffering from a disease or undergoing a form of treatment which can be expected to influence immunological functions
* Suffering from a chronic, degenerative and/or inflammatory disease of the central nervous system
* HIV-positivity (no special HIV test required for the purpose of the study)
* Suffering from a febrile disease
* History of vaccination against yellow fever and/or Japanese encephalitis
* Participation in another clinical trial

Ages: 6 Months to 47 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Dates: Start 1998-04; Study Completion 1999-06

CONTACTS AND LOCATIONS:
Overall Officials: Baxter BioScience Investigator, Principal Investigator — Baxter Healthcare Corporation
Locations (7):
- Austria (7):
  - Wiener Strasse 50/2, Kapfenberg
  - Erzherzog Johann Strasse 9, Leoben
  - Fronleichnamsweg 10, Liezen
  - Hauptstrasse 61, Linz
  - Brauhausgasse 1, Mürzzuschlag
  - Conrad-von-Hötzendorf Strasse, Voitsberg
  - Grieskirchner Strasse 17, Wels